CLINICAL TRIAL: NCT03932916
Title: Evaluation of Safety and Pharmacokinetic Profiles of a Single-dose HHT201 in Healthy Subjects
Brief Title: Safety and Pharmacokinetic of Donepezil Pamoate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Synergy Pharmaceutical Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DON101-CTP
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: AD
MeSH Terms: interventions — Injections; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group 1 (Experimental): HHT201 17mg injection
  Interventions: Drug: Donepezil Pamoate for Injection 17mg
- experimental group 2 (Experimental): HHT201 34mg injection
  Interventions: Drug: Donepezil Pamoate for Injection 34mg
- experimental group 3 (Active Comparator): Donepezil Hydrochloride oral tablet 5mg
  Interventions: Drug: Donepezil Hydrochloride 5mg

INTERVENTIONS:
Drug: Donepezil Pamoate for Injection 17mg — A dosage of 17mg HHT201 will be injected into the muscle in the gluteus once.
  Other Names: HHT201
  Arms: experimental group 1
Drug: Donepezil Pamoate for Injection 34mg — A dosage of 34mg HHT201 will be injected into the muscle in the gluteus once.
  Other Names: HHT201
  Arms: experimental group 2
Drug: Donepezil Hydrochloride 5mg — A tablet of 5mg Donepezil Hydrochloride will be administered once.
  Other Names: Aricept
  Arms: experimental group 3

SUMMARY:
The objective of this study is to evaluate the safety and pharmacokinetic profiles of HHT201 in healthy subjects.

DETAILED DESCRIPTION:
The study aims to evaluate the safety, pharmacokinetics and to determine the potential dose limiting toxicity of HHT201 in healthy subjects between the ages of 20-59, 6 in 17mg dose group and 20 in 34mg dose group. Another 12 subjects will be administered a tablet of 5mg Donepezil Hydrochloride to get the PK profile of Donepezil as reference. Eligible subjects will be accepted into the protocol after review and providing voluntary written informed consent forms and completion of a comprehensive medical, physical examination, and routine laboratory assessment.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy subjects, male or female
* between the ages of 20 and 60 years
* A body mass index (BMI), calculated as weight in kg/(height in m)², from 19 to 28 kg/m², and female weight≥45kg, male weight≥50kg
* Able to provide written informed consent forms

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders
2. Resting pulse rate <55/min or >100/min; Sitting systolic blood pressure <90mmHg or >140mmHg, diastolic blood pressure <60mmHg or >90mmHg
3. ALT or Cr, BUN exceeding the upper limit of normal value; test results of urine protein was "++"
4. Clinically significant ECG abnormalities in screening or baseline, such as male QTc interval ≥450ms and female QTc interval ≥470ms, and were considered inappropriate for inclusion by the researchers
5. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody
6. History or presence of drug or alcohol abuse
7. Positive pregnancy test result, or plan to be pregnant if female
8. An unwillingness or inability to comply with food and beverage restrictions within 24 hours prior to dosing
9. Participation in any other investigational drug trial within 30 days prior to screening.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Cmax of Donepezil | Blood samples collected over a 35 days period
  Maximum observed concentration of drug substance in plasma.
Tmax of Donepezil | Blood samples collected over a 35 days period
  Time when the maximum concentration is acheived
AUClast of Donepezil | Blood samples collected over a 35 days period
  Area under the concentration-time curve from time zero to time of last measurable concentration.
AUC0-∞ of Donepezil | Blood samples collected over a 35 days period
  Area under the concentration-time curve from time zero to infinity.
t1/2 of Donepezil | Blood samples collected over a 35 days period
  The time when the concentraion of the drug eliminated to half of the initial.

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai mental health center, Shanghai, Shanghai Municipality, China